CLINICAL TRIAL: NCT04753190
Title: Adolescent Circadian Phase Shifts: Novel Time-of-day Targets for Bright Light
Brief Title: Light Timing Study
Acronym: ALT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: R01HL151512 (NIH)
Record Dates: First submitted 2021-02-08; First posted 2021-02-15 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Chronobiology; Light; Sleep; Circadian Rhythm; Adolescence
Keywords: Sleep; Circadian Rhythm; Adolescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dim Room Light Control (Placebo Comparator): Participants in the dim room light control group will not receive any bright light exposure.
  Interventions: Behavioral: Baseline Sleep Satiation and Phase Stabilization; Behavioral: Gradually Shifted Sleep
- Morning Bright Light Only (MBL) (Experimental): Participants in the morning bright light (MBL) group will receive a 3-h bright light exposure from 2 light boxes on 3 consecutive mornings in the laboratory. Bright light will be timed for each individual based on their baseline sleep schedule to shift the circadian timing system earlier ("phase advance").
  Interventions: Behavioral: Baseline Sleep Satiation and Phase Stabilization; Behavioral: Gradually Shifted Sleep
- Afternoon Light Only (ABL) (Experimental): Participants in the afternoon bright light (ABL) group will receive a 3-h bright light exposure from 2 light boxes on 3 consecutive afternoons in the laboratory. Bright light will be timed for each individual based on their baseline sleep schedule to shift the circadian timing system earlier ("phase advance").
  Interventions: Behavioral: Baseline Sleep Satiation and Phase Stabilization; Behavioral: Gradually Shifted Sleep
- Morning + Afternoon Light (MBL+ ABL) (Experimental): Participants in the morning bright light + afternoon bright light (MBL+ ABL) group will receive bright light from 2 light boxes on 3 consecutive days in the laboratory. The morning exposure will be 1.5 h and the afternoon exposure will be 1.5 h. Bright light exposures will be timed for each individual based on their baseline sleep schedule to shift the circadian timing system earlier ("phase advance").
  Interventions: Behavioral: Baseline Sleep Satiation and Phase Stabilization; Behavioral: Gradually Shifted Sleep

INTERVENTIONS:
Behavioral: Baseline Sleep Satiation and Phase Stabilization — All participants will be assigned a 9-h sleep opportunity for the first week of the 2-week study. This will ensure that adolescents are not sleep restricted before living in the laboratory during the second week of the study. The 9-h sleep schedule will be individually timed from his/her averaged wake time (± 15 mins) before the study begins. Assigned bedtime will be 9 h before wake.
Behavioral: Gradually Shifted Sleep — For all participants, their assigned baseline sleep/wake schedule will gradually shift earlier over 3 days in the laboratory to facilitate the phase advance shift of the circadian system.

SUMMARY:
Chronic circadian misalignment and sleep restriction peak during late adolescence, and are associated with morning daytime sleepiness, poor academic performance, conduct problems, depressed mood, suicidal ideation, substance use, insulin resistance, and obesity. Bright light exposure from light boxes can shift rhythms earlier (phase advance) to facilitate earlier sleep onset and reduce morning circadian misalignment and the associated risks. To phase advance circadian rhythms, the investigators' PRCs showed that the ideal time to begin light exposure was slightly before wake-up time and light should be avoided around bedtime because this is when light produces maximum phase delay shifts. An unexpected finding from these results, however, was a second advancing region in the afternoon (~6 to 9 h after habitual wake-up time) suggesting that afternoon light may have more circadian phase advancing ability than traditionally thought. The overall goal of this mechanistic study is to follow-up on the unexpected PRC findings and test whether individually-timed afternoon light alone and in combination with morning bright light can shift circadian rhythms earlier in older adolescents. Four groups will be compared in a randomized parallel group design: afternoon bright light, morning bright light, morning + afternoon bright light, and a dim room light control. Adolescents will complete a 2-week protocol. After a baseline week with a stable sleep schedule, adolescents will live in the laboratory for 7 days. Sleep/dark and the time of bright light exposure will gradually shift earlier. Bright light (~5000 lux) will be timed individually based on his/her stable baseline sleep schedule. The first 3-h morning bright light exposure will begin 1 h before wake on the first morning. The first 3-h afternoon bright light exposure will begin 5 h after wake. The morning + afternoon exposures will begin at the same times, but each exposure will be 1.5 h so that a total of 3 h of bright light per day will be given to each group except the dim light control group. Phase shifts of the circadian clocks marked by the dim light melatonin onset (DLMO) is the main outcome. Investigators hypothesize that afternoon bright light will work synergistically with morning bright light to produce larger shifts than morning or afternoon bright light alone. These data could challenge the current understanding of how to use bright light to shift circadian rhythms earlier.

DETAILED DESCRIPTION:
Participants will complete a 14-day protocol. On days 1-7, participants will sleep at home on a stable sleep schedule that requires 9 h of time in bed in the dark. This will ensure that participants are not sleep deprived before beginning the lab sessions. Wake time will be the average of the self-reported wake-up time (± 15 mins) before the study begins measured from pre-study sleep logs collected for a week or more. Bedtime will be 9 h before wake-up time. A device worn on the wrist that measures activity (actigraph), sleep diaries, and daily telephone messages will monitor compliance to the sleep schedule. Participants will visit the lab at least once during this week to download and review their data. If participants are not compliant to the sleep schedule, they will be dropped from the study.

On days 8-13, participants will live in the laboratory for seven days. On day 8, participants will arrive at the laboratory in the afternoon, and shortly after, will begin a baseline circadian phase assessment to determine baseline dim light melatonin onset (DLMO), a reliable marker of the circadian timing system. On day 9, participants will sleep on their stable 9-h sleep schedule in the laboratory. Their 9-h fixed sleep schedule will be shifted by 1 h per day over 3 days. Participants will sleep in dark bedrooms in the lab. During scheduled wake, participants will remain awake in normal dim room light except during bright light sessions, when light will range from 5000 to 7000 lux. Study groups will differ by the light exposure they receive during the lab sessions. In the afternoon bright light (ABL) group, participants will be exposed to 3 h of bright light on 3 consecutive afternoons. On the first day (day 10), light boxes will be turned on 5 h after fixed wake-up time. Then, the start of the light exposure will move 1 h earlier each day. In the morning bright light (MBL) group, participants will be exposed to 3 consecutive mornings of 3 h of bright light. On the morning of day 11, the 3-h bright light exposure will begin 1 h before their stable wake-up time. In the morning + afternoon bright light (MBL + ABL) group, bright light will begin at the same times as the ABL and MBL groups and participants will received the same duration of bright light per day (3 h) as the ABL and MBL groups because the duration of each exposure will be 1.5 h instead of 3 h. Both bright light exposures will move 1 h earlier on subsequent days. In the room light control group, participants will complete the same 7-day lab session, except remain in dim room lighting. All participants will complete a final circadian phase assessment at the end of the 7-day lab session (day 13).

ELIGIBILITY:
Inclusion Criteria:

* between 18-20 years old
* lives in or near Chicago, IL

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 113 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Dim Light Melatonin Onset (DLMO) Phase Shift Change | Change in DLMO phase from baseline (day 8) to final phase assessment (day 13)
  Saliva sampling for the baseline DLMO will begin 6 hours before baseline bedtime and end 2 hours after baseline bedtime to capture the rise of endogenous melatonin. Sampling for the final DLMO will begin 7 hours before baseline bedtime and end 2 hours after baseline bedtime. Participants remain awake and seated in comfortable recliners in dim light (< 5 lux), except when they need to use the adjoining restroom (also < 5 lux). Saliva samples are collected every 30 minutes using Salivettes, The samples are immediately centrifuged and frozen, and later shipped on dry ice to SolidPhase, Inc. (Portland, ME), where they are analyzed for melatonin using direct radioimmunoassay (RIA). We compute the DLMO using a 4 pg/mL threshold; the time at which melatonin values surpass this threshold is the DLMO. Baseline - Final DLMO will define the phase shift change of the central circadian clock.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States